CLINICAL TRIAL: NCT03390088
Title: The Clinical Profiles and Treatment Management of Chronic Heart Failure in Azerbaijan
Brief Title: Heart Failure Management in Azerbaijan
Acronym: CHF-AZ
Status: Withdrawn | Type: Observational
Why Stopped: The estimated number of patients could not be recorded in this study
Sponsor: Prof. Dr. Mehdi Zoghi (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Mehdi Zoghi, President of WHFS, World Heart Failure Society
Organization: World Heart Failure Society (Other)
Other Study IDs: 2018-1
Record Dates: First submitted 2017-12-26; First posted 2018-01-04 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Heart Failure
Keywords: Heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is proposed to determined a national database of the etiologies, clinical and the demographic profile, using diagnostic tests and treatment of outpatients with chronic heart failure in Azerbaijan population.

DETAILED DESCRIPTION:
Chronic heart failure remains the leading cause of hospitalization for those over the age of 65 and expected to increase over the next 25 years with advancing life span. Being a progressive syndrome, CHF decreases the quality of life and place an economic burden on health care system.

Advanced technologies in interventional cardiology, better organization of angiographic laboratories and primary prevention of coronary artery disease as the leading cause of HF, allowed warning its development in CAD patients. But the incidence and prevalence of CHF continue to increase with age as heart failure with preserved ejection fraction predominates in elderly patients. For the moment more than 23 million people over the world suffer from heart failure.

The prevalence of these patients remains very high even in USA - over 5.8 million.However, there is no any database for heart failure patient in Azerbaijan.The purpose of this study is to compose a national database of the etiologies, clinical and demographic characteristics, using diagnostic tests and management of outpatients heart failure in Azerbaijan population.

ELIGIBILITY:
Inclusion :

* Patients >18 years olds
* Clinical diagnosis of heart failure
* NYHA class II-IV heart failure

Exclusion :

* Patients <18 years old
* Failure to obtain informed consent
* Pregnant or lactating

Previous cardiac transplantation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: outpatients with chronic heart failure
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-01-28 (Actual); Primary Completion 2019-12-28 (Estimated); Study Completion 2020-01-14 (Estimated)

PRIMARY OUTCOMES:
Heart failure related hospitalization | 6 months
  Heart failure related hospitalization within 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Yasmin Rustamova, Baku, Azerbaijan